CLINICAL TRIAL: NCT03595696
Title: Effect of a Core Strengthening Program on Diastasis Rectus Abdominus in Postpartum Women
Brief Title: Core Strengthening for DRA in Postpartum Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2017-1999
Record Dates: First submitted 2018-07-11; First posted 2018-07-23 (Actual); Last update posted 2019-11-20 (Actual); Status verified 2019-11

CONDITIONS: Diastasis Recti; Postpartum; Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Core Strengthening Exercise Intervention (Experimental): All subjects will participate in the study for a total of 24 consecutive weeks. During the first 12 weeks, subjects will participate in weekly online exercise classes for Core Muscle Strength training and will be asked to perform daily homework assignments. Following completion of the 12-week intervention, subjects will be asked to continue the exercises on their own.
  Interventions: Other: Core Muscle Strength Training
- Control+Core Strengthening Exercise (Active Comparator): All subjects will participate in the study for a total of 24 weeks. During the first 12 weeks, subjects will serve as the control group, and they will be advised to continue their baseline level of exercise and lifestyle. During the subsequent 12 weeks, subjects will participate in the exact same program as Group A performed during the first 12 weeks (Core Muscle Strength Training).
  Interventions: Other: Core Muscle Strength Training

INTERVENTIONS:
Other: Core Muscle Strength Training — Targeted weekly workouts consisting of low-impact aerobic exercises and resistance exercises designed to address muscle imbalance common in women who exhibit DRA and to prompt automatic core engagement while performing compound, multi-joint movements.

SUMMARY:
This study will prospectively measure the effectiveness of a core strengthening program on reducing the inter-rectus distance (IRD) and abdominal wall muscle contraction in postpartum women with diastasis rectus abdominus (DRA). Additionally, this study will aim to investigate and clarify the association between IRD and low back pain.

DETAILED DESCRIPTION:
DRA is a separation of the abdominal wall muscles that commonly occurs during pregnancy and is caused by the stretching of the linea alba to accommodate a growing fetus. Separation of core muscles is thought to be factor in postpartum low back pain, stress urinary incontinence, and core strength, as well as being cosmetically undesirable. This study will evaluate the effect of a core strengthening program on shortening the IRD and improving the connectivity and strength of abdominal wall muscles in postpartum women with a DRA. It will also investigate the relationship between IRD and low back pain.

ELIGIBILITY:
Inclusion Criteria:

* Healthy women who have given birth within the last 36 months but are at least 12 weeks postpartum
* Not currently pregnant
* Current DRA diagnosed using ultrasound with an IRD of at least 2.0 cm

Exclusion Criteria:

* History of ventral/umbilical hernia prior to pregnancy
* >36 months postpartum
* Currently pregnant
* Beighton's score >5/9
* Unable to participate in a regular core strengthening program
* Unable to attend the three data collection sessions

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-07-16 (Actual); Study Completion 2019-07-16 (Actual)

PRIMARY OUTCOMES:
Change in inter-recti distance (IRD) | Up to 24 weeks
  Change in IRD will be measured using palpation and musculoskeletal ultrasound.

SECONDARY OUTCOMES:
Abdominal wall muscle function | Up to 24 weeks
  Measured using musculoskeletal ultrasound at rest and during contraction (abdominal draw-in maneuver).
Low back pain | Up to 24 weeks
  Measured using the Quebec Back Pain Disability Scale. Scores range from 0 to 100, with 100 representing higher disability.
Pelvic function | Up to 24 weeks
  Measured using the Pelvic Organ Prolapse/Urinary Incontinence Sexual Function. Scores range from 0 to 48, with a higher score representing greater impairment.
Stress urinary incontinence | Up to 24 weeks
  Measured using the International Consultation on Incontinence Modular Questionnaire-Urinary Incontinence Short Form. Scores range from 0 to 21, with higher scores indicating increased severity.
Body image | Up to 24 weeks
  Measured using the Body Shape Questionnaire. Scores range from 16 to 96, with a higher score representing impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Ellen Casey, MD, Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- Hospital for Special Surgery, New York, New York, United States